## ENCOURAGE APP – statistical analysis plan:

For the primary outcome, a one-way repeated measures ANOVA or Mann-Whitney Test will be used to examine changes in the number of breaks in sedentary time from baseline to 1-month, depending if the data are normally distributed.

Other secondary, continuous outcome measures will be analyzed with a one-way repeated measures ANOVA or Mann-Whitney Test from baseline to 1 week, 1-month, 2-month, 3-month, 4-month, 5-month, and 6-month depending if the data are normally distributed. Categorical variables will be compared using a Chi-Square test. Relationships between variables will be assessed using Pearson or Spearmen correlations, as well as multivariable linear or logistic regression.